CLINICAL TRIAL: NCT06695715
Title: Effect of Heart Rate Variability Biofeedback, Interoceptive Training, and Mindfulness on Stress Reduction in the University of Seville Academic Community (Faculty, Administrative Staff, and Students)
Brief Title: Effects of HRV Biofeedback, Interoceptive Training, and Mindfulness on Stress in University Students and Staff
Acronym: BIMStress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Francisco M. Ocaña Campos, PhD. Associate Professor of Psychobiology. Principal Investigator of the Wellness Neuroscience Group-, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SICEIA-2024-002431
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Stress; Anxiety
Keywords: Stress; Anxiety; Mindfulness; HRV Biofeedback; qEEG; University Students and Staff; Interoception
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mindfulness (Experimental): The Mindfulness Training program will be based on the Mindfulness-Based Stress Reduction (MBSR) program and Jon Kabat-Zinn's Mindful Awareness practices, but will also include elements of self-compassion and acceptance.
  Intervention: During the six weeks of the program, participants will take part in a guided 45-minute formal session. Examples of formal guided meditations include mindfulness of breath and mindfulness of thoughts, feelings, and physiological sensations. Informal meditation practices will consist of brief pauses throughout the day, during which participants will voluntarily direct their attention to the present moment without judgment. Finally, participants will be provided with 10 audio recordings of guided meditations, recorded by a member of the research team, to support formal meditation at home (10-15 minutes four times a week), as well as a series of readings focused on the concepts of acceptance and self-compassion.
  Interventions: Behavioral: Mindfulness Training Program
- HRV Biofeedback Training (HRV-BF) (Experimental): The HRV BF training will last for 6 weeks. There will be five training sessions per week, including four home sessions and one in-person session at the Neurociencia del Bienestar group laboratory (CTS-1129) at the Faculty of Psychology of the University of Seville. Each session will last 20 minutes. The laboratory session will be conducted using the Procomp Infiniti biofeedback equipment (Thought Technologies). For the home HRV-BF sessions, we will use a novel methodology recently described (Schumann et al., 2021). The heart rate will be recorded using a sensor embedded in a strap that will be worn around the participant's chest (H10/H7 heart rate sensor; Polar Electro Oy, Kempele, Finland). Via Bluetooth, the mobile app EliteHRV (Elite HRV LLC, 2017) will collect data from the sensor, store the recordings, and display the heart rate. The heart rate oscillations will be shown on the participants' smartphone screens as real-time visual feedback of their heart rate.
  Interventions: Behavioral: HRV Biofeedback
- Interoceptive Training (Experimental): During the 6 weeks of the program, participants in this group will complete a 45-minute formal guided interoceptive training session at the Faculty of Psychology. During these sessions, the focus will be on developing internal body awareness through various strategies. Participants will learn to pay attention to internal sensations such as breathing and muscle tension using guided techniques. The program will include exercises to feel the flow of breath and relax specific areas of the body. The trainer will provide feedback and adjust techniques based on the participants' needs. Instructions will be given on how to integrate these practices into daily life to improve self-care and self-regulation. Finally, participants will be provided with 10 audio recordings of guided interoceptive exercises, recorded by a member of the research team, to support formal training at home (10-15 minutes, four times a week).
  Interventions: Behavioral: Interoception Training
- Waiting list control group (No Intervention): Participants assigned to the waitlist control group will be key to ensuring the validity and reliability of the results of this project, allowing for precise and controlled comparisons of the effectiveness of the different training programs. These participants will also be evaluated at the beggining and the end, even though they will not participate in any training program. Once the program is completed, they will be offered the opportunity to participate in some of the training programs used in this project.

INTERVENTIONS:
Behavioral: Mindfulness Training Program — This mindfulness training program is based on the Mindfulness-Based Stress Reduction (MBSR) model developed by Jon Kabat-Zinn, incorporating elements of self-compassion and acceptance. What sets this program apart is its integration of both formal and informal practices. Participants engage in 45-minute guided sessions focused on breath awareness and the observation of thoughts, emotions, and physical sensations. Additionally, informal practices include brief daily moments of present-moment awareness. Participants will also receive 10 audio recordings for at-home practice, enhancing the program's accessibility and supporting consistency.
  Arms: Mindfulness
Behavioral: HRV Biofeedback — This HRV biofeedback training program is distinguished by its combination of advanced technology and a novel at-home methodology. Participants will engage in five weekly sessions, with four conducted at home using a heart rate sensor and the EliteHRV mobile app, which provides real-time feedback on heart rate variability. One session per week will take place in the lab, utilizing the Procomp Infiniti biofeedback system. The at-home approach is based on recent research (Schumann et al., 2021), offering participants a flexible yet structured method to practice biofeedback and improve heart rate variability over the six-week program.
  Arms: HRV Biofeedback Training (HRV-BF)
Behavioral: Interoception Training — The interoception training program stands out by its focus on developing internal body awareness through structured guided sessions. Participants will engage in weekly 45-minute formal sessions at the university, where they will learn to focus on internal sensations like breath and muscle tension using specific techniques. Additionally, participants will receive 10 guided interoceptive exercises to practice at home, four times a week. This program not only focuses on the physical sensations but also integrates these practices into daily life, aiming to improve self-care and self-regulation over the six weeks, with personalized feedback provided.
  Arms: Interoceptive Training

SUMMARY:
The goal of this clinical trial is to learn if Heart Rate Variability Biofeedback (HRV-BF), Mindfulness programs, and Interoception training can reduce stress, improve well-being, and induce brain changes in university students and staff at the University of Seville. The main questions it aims to answer are:

* Does HRV-BF training reduce stress, improve emotional regulation, and cause measurable brain changes in participants?
* Does Mindfulness training reduce perceived stress, improve mental health, and lead to changes in brain activity?
* Does Interoception training enhance emotional self-regulation, reduce stress, and produce changes in brain function?
* How do the effects on the brain compare between the different types of training (HRV-BF, Mindfulness, and Interoception)?

If there is a comparison group: Researchers will compare participants who receive HRV-BF, Mindfulness, and Interoception training to a waitlist control group to see if any of these interventions lead to greater reductions in stress, improvement in emotional regulation, or brain activity changes.

Participants will:

* Complete pre- and post-training assessments to measure stress levels, anxiety, emotional regulation, and brain activity using EEG (electroencephalography).
* Participate in one of three interventions:

HRV-BF training, where participants learn to use biofeedback to improve heart rate variability and manage stress.

Mindfulness-based stress reduction, which involves meditation and mindful awareness techniques to reduce stress and improve mental health.

Interoception training, where participants learn to focus on internal bodily signals (like heartbeat and breath) to improve emotional regulation and manage stress.

Each intervention will last six weeks, and participants will be assessed at the beginning and end of the program. This study aims to determine which intervention is most effective at reducing stress, improving mental health, and producing beneficial changes in brain activity in university community members.

DETAILED DESCRIPTION:
All people experience stress at certain times, as it is a natural response to threats. However, a complex interaction of social, technological, work-related, and environmental factors has contributed to a prolonged stress response, leading to a rise in chronic anxiety problems throughout the 21st century. According to the National Health Survey, 6.7% of adults report chronic anxiety. Furthermore, there is a significant gender gap, with prevalence being twice as high in women as in men (9.1% in women and 4.3% in men). Members of the university community are not immune to this issue. Several recent studies have highlighted that, for example, university students are exposed to alarmingly high levels of stress. According to various surveys, 35% of higher education students suffer from anxiety, and 30% suffer from depression. Moreover, this is a global phenomenon. In the United States, a survey by the American College Health Association shows that stress has become the most serious obstacle to studying among American students; in the United Kingdom, another study shows that 45% of students report feeling stressed by their courses. Gender, as a demographic factor, also seems to play a significant role, as female students are the most affected, not only by stress but also by other aspects of mental health. In fact, this represents another problem: most university students report, in addition to stress, a large number of symptoms associated with mental health problems, such as sadness, lack of energy or motivation, anxiety, depression, hopelessness, insomnia, irritability, mood swings, panic, or self-harm ideations. Another aspect that has negatively impacted not only stress but also the mental health of the student population worldwide has been the COVID-19 pandemic. Several studies have shown an increase in stress among university students from various countries, both European and non-European, following the start of the pandemic. Regarding the working members of the university community, such as teaching and research staff (PDI) or administrative and service staff (PTGAS), chronic work-related stress and associated pathologies, such as burnout syndrome, are among the leading emerging psychosocial risks. In this population, sociodemographic factors such as age and gender play a fundamental role, with younger staff and, within this group, women, scoring the highest in areas related to emotional exhaustion and stress. In particular, among the PDI, younger women in the social sciences, in the early stages of their professional development, with lower contractual figures and high teaching loads, experience higher levels of stress. Both stress and other mental health issues decrease quality of life, increase absenteeism among workers and students, and reduce professional and academic performance within the university community. Therefore, the development of preventive and palliative strategies, within the university itself, to reduce the impact of stress and protect the health and well-being of its members is highly recommended. By implementing these measures and promoting a culture of well-being, universities can help mitigate the negative impact of stress and improve the quality of life of their community members. In this context, it is a priority to develop new, cost-effective, and accessible stress reduction programs within the university space. Three approaches that meet these criteria are Heart Rate Variability Biofeedback (HRV-BF), Mindfulness-based programs (MBPs), and Interoception Training programs (ITPs). Heart Rate Variability (HRV) is the temporal variation between successive heartbeats (RR intervals) and serves as a quantitative biomarker of the autonomic nervous system (ANS) balance and physiological stress. Dysregulation of the ANS, mainly increased sympathetic activity and decreased parasympathetic activity (vagal hypofunction), is a common feature of chronic stress, anxiety, and mood disorders and appears to be a central biological substrate linking these disorders to a range of physical dysfunctions. Alterations in the functioning of the autonomic nervous system that promote a decrease in vagal (parasympathetic) activity are reflected in reductions in HRV indices, which in turn are associated with emotional dysregulation, decreased psychological flexibility, and faulty social engagement-disorders linked to hypoactivity in the prefrontal cortex. Similarly, work-related stress has been shown to reduce HRV. On the other hand, high HRV indicates greater parasympathetic activity and better self-regulation, which is associated with a lower cardiovascular risk and better cognitive performance. Together, these findings support the idea that HRV could represent a useful endophenotype for psychological/physical comorbidities, and its measurement and routine application should be recommended to assess the effectiveness of training based on these measures for emotional regulation dysfunctions. Indeed, HRV is currently considered a biomarker of the ANS function associated with both physical and mental health and well-being. Biofeedback is a way of helping individuals develop greater awareness and the ability to regulate their physiological functioning using signals from their own bodies to improve their well-being, health, and performance. Specifically, HRV biofeedback is a well-established and empirically supported technique to improve emotional self-regulation and alleviate symptoms of stress, anxiety, and other psychophysiological disorders. Quantitative studies suggest that HRV-BF training reduces anxiety by 26%, fatigue by 15%, blood pressure by 10%, cholesterol by 14%, and increases fitness levels by 40%. During HRV-BF training, individuals learn to breathe slowly, gradually reaching the optimal breathing frequency that maximizes HRV. Additionally, it has recently been shown that this training induces plastic changes in brain activity and connectivity in regions related to emotion regulation and executive functions. Although there are numerous studies highlighting the effectiveness of HRV-BF in reducing stress, most of them rely on subjective measures obtained through self-reports, so there is a need for research that includes both neuropsychological and physiological parameters when analyzing the effectiveness of biofeedback training in preventing and reducing stress in high-demand work or academic environments. Mindfulness has been defined as "paying attention in a particular way, on purpose, in the present moment, and without judgment". The first mindfulness-based stress reduction (MBSR) program was developed over 50 years ago by Jon Kabat-Zinn, and since then, countless scientific studies have demonstrated the effectiveness of MBPs in reducing stress, as well as their efficacy in treating anxiety and depression disorders. In fact, a recent randomized clinical trial has shown that MBPs are as effective as escitalopram (first-choice medication) in treating anxiety disorders. Various formats of MBPs for stress reduction among university community members have been used in several studies, varying primarily in the focus of attention, duration, or the traditional in-person nature of the training versus those guided by new technologies (apps). Despite this variability, all these studies show a positive effect of these programs on perceived stress in this population. Also, like HRV-BF, all reviewed studies rely on self-reports of stress without measuring or evaluating any psychophysiological or neurophysiological parameters (objective). In conclusion, the success of MBPs in reducing or mitigating stress in university community members makes these techniques a useful tool for preventing psychosocial risks, such as stress, in university settings. In recent years, our understanding of the physiological changes associated with mindfulness practice, as well as the potential mechanisms underlying its efficacy and effectiveness as a treatment for various mental disorders, has significantly advanced. For example, it is widely accepted that the implementation of an MBP in non-clinical samples leads to an increase in HRV. On the other hand, similarly to the case of HRV-BF, mindfulness practice can modulate prefrontal cortex activity, promoting emotional regulation, cognitive control, attentional stability, and resilience to stress. These changes may underlie many of the cognitive and emotional benefits associated with mindfulness training. However, individual responses to mindfulness practices can vary, and further research is needed to fully understand the underlying mechanisms of these effects. Interoception is the process by which the nervous system perceives, interprets, and integrates signals from within the body, including sensations from internal organs and physiological states. This encompasses sensory signaling (neural and humoral), perceptual processing, and the psychological representation of such sensations. In simpler terms, interoception is the ability to feel and understand what is happening inside the body, such as heartbeat, breathing, hunger or fullness, thirst, and body temperature. Interoception plays a key role in emotion regulation, decision-making, self-awareness, and health regulation. Some authors suggest that interoception plays a key role in emotional experience, as it allows individuals to recognize their emotional states and regulate them. It has also been shown that emotional dysregulation can result in distorted perceptions of interoceptive information, and vice versa, that training interoception improves emotional regulation and helps reduce anxiet. In fact, recent studies have shown that interoception training can improve mental health outcomes, including emotional regulation and stress management, and it is considered a promising intervention for those suffering from high levels of stress and anxiety. Recent research into interoception has led to the development of interoceptive training programs, which have proven effective in reducing stress, improving emotion regulation, and increasing mindfulness. A growing body of evidence suggests that ITPs can enhance emotional awareness and regulation and improve autonomic nervous system regulation, potentially contributing to reduced anxiety and stress. To summarize, interoception-based interventions provide promising strategies for reducing stress and improving well-being by fostering greater body awareness and self-regulation. Like HRV-BF and MBPs, ITPs can be easily implemented in university settings and may represent a cost-effective alternative for managing stress. However, like mindfulness, it would benefit from more research into the neurophysiological and cognitive effects of such training, especially in terms of potential changes in brain activity related to emotional regulation and stress reduction.

Although the scientific evidence on the benefits of HRV-BF (Heart Rate Variability Biofeedback), MBPs (Mindfulness-Based Programs), and ITPs (Interoception Training Programs) in relation to stress reduction is more than notable, to the best of our knowledge, there are no randomized experimental studies analyzing the effectiveness of HRV-BF, MBPs, and ITPs in the prevention and/or reduction of stress that rely on the evaluation of variables of different natures: psychological, neuropsychological, psychophysiological, and neurophysiological. Furthermore, it would be of great interest to conduct a long-term evaluation of the effects of these training programs.

The aim of this project is to analyze the impact of a HRV-BF training program, an MBP, and an ITP among members of the University of Seville community, evaluating their effects on stress in both women and men through neuropsychological, psychophysiological, and brain activity measures.

ELIGIBILITY:
Inclusion Criteria:

* Members of the University of Seville community over 18 years old (students, teaching staff, and administration and service staff)
* Be able to attend at least five of the six weeks of the Heart Rate Variability Biofeedback (HRV-BF) and Mindfulness (PEM) training programs
* Have a smartphone.

Exclusion Criteria:

* Members of the University of Seville community who are experiencing severe anxiety or depression; a serious mental illness, such as hypomania or psychotic episodes; recent grief or a major loss; any heart disease; any other serious physical or mental health condition that may affect their ability to participate in the training program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  We measure stress using the Spanish Version (2.0) of the Perceived Stress Scale (PSS). Authors: Cohen S, Kamarck T, Mermelstein R. (1983); adapted by Eduardo Remor (2001). Validation data: Remor E, Carrobles JA. (2001). Spanish Version of the Perceived Stress Scale (PSS-14): Psychometric Study in an HIV+ Sample. Ansiedad y Estrés, 7 (2-3), 195-201. // Remor E. (2006). Psychometric Properties of a European Spanish Version of the Perceived Stress Scale (PSS). The Spanish Journal of Psychology, 9 (1), 86-93.
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  HRV analysis in time domain
  - SDNN (Standard Deviation of NN intervals): represents overall HRV and total autonomic activity. Units: ms.
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  HRV analysis in time domain
  - RMSSD (Root Mean Square of Successive Differences): reflects parasympathetic (vagal) activity. Units: ms
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  HRV analysis in time domain
  - NN50 / pNN50 (Number or percentage of consecutive NN intervals differing by >50 ms): indicates short-term vagal regulation. Units: %
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  HRV analysis in Frequency-Domain
  - Total Power (0-0.4 Hz): Overall HRV across all frequency bands. Units: ms².
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  HRV analysis in Frequency-Domain
  - HF (High Frequency, 0.15-0.4 Hz): Reflects parasympathetic activity (vagal tone). Units: ms²
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  HRV analysis in Frequency-Domain
  - LF (Low Frequency, 0.04-0.15 Hz): Represents a mix of sympathetic and parasympathetic activity. Units: ms².
Heart Rate Variability (HRV) as a biomarker of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  HRV analysis in Frequency-Domain LF/HF Ratio: Balance between sympathetic and parasympathetic activity. Units: ms².
QEEG as a biomarker of Stress. Frequency Bands and Power Analysis | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  Delta Power (0.5-4 Hz).Units: Microvolts squared (µV²) or decibels (dB).
  Theta Power (4-8 Hz). Units: µV² or dB.
  Alpha Power (8-12 Hz). Units: µV² or dB.
  Beta Power (12-30 Hz). Units: µV² or dB.
  Gamma Power (>30 Hz). Units: µV² or dB.
QEEG as a biomarker of Stress. Ratios as Indicators of Stress | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  Theta/Beta Ratio: Evaluates emotional regulation and attentional processes. Stress relevance: High ratios often reflect underarousal or emotional stress, while low ratios suggest hyperarousal or anxiety.
  Alpha/Theta Ratio: Indicates balance between relaxation and alertness. Stress relevance: Lower ratios suggest stress or difficulty in maintaining relaxed alertness.
  Alpha/Beta Ratio: Reflects relaxation versus stress or anxiety levels. Stress relevance: Low ratios are associated with stress or hyperactivity.
QEEG as a biomarker of Stress. Coherence Measures | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  Coherence (between regions): Measures synchronization between two brain areas. Units: Dimensionless (0-1).
  Stress relevance: High coherence may indicate rigid patterns (hyperconnectivity) due to stress, while low coherence may indicate disconnection or poor integration.
QEEG as a biomarker of Stress. Connectivity Measures | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  Phase Lag Index (PLI): Quantifies the phase relationship between EEG signals, indicating functional connectivity. Units: Dimensionless (0-1).
  Stress relevance: Abnormal PLI values (too high or too low) may reflect stress-induced connectivity changes.
QEEG as a biomarker of Stress. Asymmetry Measures | Baseline or pretraining (one week before training programs) and posttraining (one week after training programs; 7 weeks after first measure)
  Frontal Alpha Asymmetry:
  Compares alpha power between left and right frontal lobes (F3-F4). Units: Log-transformed ratios (e.g., log(left alpha) - log(right alpha)). Stress relevance: Greater right frontal alpha (reduced activity in the right hemisphere) is linked to negative affect or stress

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Ocaña, PhD, Principal Investigator — Wellness Neuroscience Group. University of Seville
Locations (1):
- Faculty Of Psychology. University of Seville, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy KJ, Menon KR, Thattil A. Academic Stress and its Sources Among University Students. Biomed Pharmacol J. 2018, 11(1).
- [Background] Marcatto F, Colautti L, Filon FL, Luis O, Di Blas L, Cavallero C, Ferrante, D. Work-related stress risk factors and health outcomes in public sector employees. Saf sci. 2016, 89, 274-278.
- [Background] Christodoulou G, Salami N, Black DS. The utility of heart rate variability in mindfulness research. Mindfulness. 2020, 11, 554-570
- [Background] Kelsey RM, Reiff S, Wiens S, Schneider TR, Mezzacappa ES, Guethlein W. The ensemble-averaged impedance cardiogram: an evaluation of scoring methods and interrater reliability. Psychophysiology. 1998 May;35(3):337-40. doi: 10.1017/s0048577298001310. PMID 9564753
- [Background] Voltmer E, Koslich-Strumann S, Walther A, Kasem M, Obst K, Kotter T. The impact of the COVID-19 pandemic on stress, mental health and coping behavior in German University students - a longitudinal study before and after the onset of the pandemic. BMC Public Health. 2021 Jul 13;21(1):1385. doi: 10.1186/s12889-021-11295-6. PMID 34256717
- [Background] Ozen NS, Ercan I, Irgil E, Sigirli D. Anxiety prevalence and affecting factors among university students. Asia Pac J Public Health. 2010 Jan;22(1):127-33. doi: 10.1177/1010539509352803. PMID 20032042
- [Background] Thayer JF, Hansen AL, Saus-Rose E, Johnsen BH. Heart rate variability, prefrontal neural function, and cognitive performance: the neurovisceral integration perspective on self-regulation, adaptation, and health. Ann Behav Med. 2009 Apr;37(2):141-53. doi: 10.1007/s12160-009-9101-z. Epub 2009 May 8. PMID 19424767
- [Background] Son C, Hegde S, Smith A, Wang X, Sasangohar F. Effects of COVID-19 on College Students' Mental Health in the United States: Interview Survey Study. J Med Internet Res. 2020 Sep 3;22(9):e21279. doi: 10.2196/21279. PMID 32805704
- [Background] Schumann A, de la Cruz F, Kohler S, Brotte L, Bar KJ. The Influence of Heart Rate Variability Biofeedback on Cardiac Regulation and Functional Brain Connectivity. Front Neurosci. 2021 Jun 29;15:691988. doi: 10.3389/fnins.2021.691988. eCollection 2021. PMID 34267625
- [Background] Paulus MP, Stein MB. An insular view of anxiety. Biol Psychiatry. 2006 Aug 15;60(4):383-7. doi: 10.1016/j.biopsych.2006.03.042. Epub 2006 Jun 14. PMID 16780813
- [Background] Maskova I. Work-related coping behaviour and experience patterns in university students: a review of 20 years of research. Front Psychol. 2023 Apr 18;14:1062749. doi: 10.3389/fpsyg.2023.1062749. eCollection 2023. PMID 37143596
- [Background] Lyzwinski LN, Caffery L, Bambling M, Edirippulige S. The Mindfulness App Trial for Weight, Weight-Related Behaviors, and Stress in University Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Apr 10;7(4):e12210. doi: 10.2196/12210. PMID 30969174
- [Background] Khalsa SS, Adolphs R, Cameron OG, Critchley HD, Davenport PW, Feinstein JS, Feusner JD, Garfinkel SN, Lane RD, Mehling WE, Meuret AE, Nemeroff CB, Oppenheimer S, Petzschner FH, Pollatos O, Rhudy JL, Schramm LP, Simmons WK, Stein MB, Stephan KE, Van den Bergh O, Van Diest I, von Leupoldt A, Paulus MP; Interoception Summit 2016 participants. Interoception and Mental Health: A Roadmap. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):501-513. doi: 10.1016/j.bpsc.2017.12.004. Epub 2017 Dec 28. PMID 29884281
- [Background] Ibrahim AK, Kelly SJ, Adams CE, Glazebrook C. A systematic review of studies of depression prevalence in university students. J Psychiatr Res. 2013 Mar;47(3):391-400. doi: 10.1016/j.jpsychires.2012.11.015. Epub 2012 Dec 20. PMID 23260171
- [Background] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569
- [Background] Hoge EA, Bui E, Mete M, Dutton MA, Baker AW, Simon NM. Mindfulness-Based Stress Reduction vs Escitalopram for the Treatment of Adults With Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Jan 1;80(1):13-21. doi: 10.1001/jamapsychiatry.2022.3679. PMID 36350591
- [Background] Gotink RA, Meijboom R, Vernooij MW, Smits M, Hunink MG. 8-week Mindfulness Based Stress Reduction induces brain changes similar to traditional long-term meditation practice - A systematic review. Brain Cogn. 2016 Oct;108:32-41. doi: 10.1016/j.bandc.2016.07.001. Epub 2016 Jul 16. PMID 27429096
- [Background] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Background] Eisenberg D, Hunt J, Speer N. Mental health in American colleges and universities: variation across student subgroups and across campuses. J Nerv Ment Dis. 2013 Jan;201(1):60-7. doi: 10.1097/NMD.0b013e31827ab077. PMID 23274298
- [Background] Eicher V, Staerkle C, Clemence A. I want to quit education: a longitudinal study of stress and optimism as predictors of school dropout intention. J Adolesc. 2014 Oct;37(7):1021-30. doi: 10.1016/j.adolescence.2014.07.007. Epub 2014 Aug 15. PMID 25128662
- [Background] Coronado-Montoya S, Levis AW, Kwakkenbos L, Steele RJ, Turner EH, Thombs BD. Reporting of Positive Results in Randomized Controlled Trials of Mindfulness-Based Mental Health Interventions. PLoS One. 2016 Apr 8;11(4):e0153220. doi: 10.1371/journal.pone.0153220. eCollection 2016. PMID 27058355
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Chandola T, Heraclides A, Kumari M. Psychophysiological biomarkers of workplace stressors. Neurosci Biobehav Rev. 2010 Sep;35(1):51-7. doi: 10.1016/j.neubiorev.2009.11.005. Epub 2009 Nov 13. PMID 19914288
- [Background] Bourion-Bedes S, Tarquinio C, Batt M, Tarquinio P, Lebreuilly R, Sorsana C, Legrand K, Rousseau H, Baumann C. Stress and associated factors among French university students under the COVID-19 lockdown: The results of the PIMS-CoV 19 study. J Affect Disord. 2021 Mar 15;283:108-114. doi: 10.1016/j.jad.2021.01.041. Epub 2021 Jan 18. PMID 33540333
- [Background] Bayram N, Bilgel N. The prevalence and socio-demographic correlations of depression, anxiety and stress among a group of university students. Soc Psychiatry Psychiatr Epidemiol. 2008 Aug;43(8):667-72. doi: 10.1007/s00127-008-0345-x. Epub 2008 Apr 8. PMID 18398558
- [Background] Aristovnik A, Kerzic D, Ravselj D, Tomazevic N, Umek L. Impacts of the Covid-19 Pandemic on Life of Higher Education Students: Global Survey Dataset from the First Wave. Data Brief. 2021 Dec;39:107659. doi: 10.1016/j.dib.2021.107659. Epub 2021 Dec 1. PMID 34869802
- [Background] Arakaki X, Arechavala RJ, Choy EH, Bautista J, Bliss B, Molloy C, Wu DA, Shimojo S, Jiang Y, Kleinman MT, Kloner RA. The connection between heart rate variability (HRV), neurological health, and cognition: A literature review. Front Neurosci. 2023 Mar 1;17:1055445. doi: 10.3389/fnins.2023.1055445. eCollection 2023. PMID 36937689